CLINICAL TRIAL: NCT03312868
Title: Phase I/II Trial of Stereotactic Body Radiotherapy for the Treatment of Solitary Bone Plasmacytoma
Brief Title: Stereotactic Body Radiotherapy for the Treatment of Solitary Bone Plasmacytoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Burocracy and funding
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Geovanne Pedro Mauro, MD, Instituto do Cancer do Estado de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 1122/17
Record Dates: First submitted 2017-10-12; First posted 2017-10-18 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Plasmacytoma
Keywords: Stereotactic Body Radiotherapy
MeSH Terms: conditions — Plasmacytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective Arm (Experimental): Prospective arm with patients being treated with SBRT
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Stereotactic Body Radiotherapy

SUMMARY:
This project aims to propose a new approach in the treatment of solitary plasmacytoma: hypofractionated irradiation alone with stereotactic technique that may contribute to the successful treatment of this disease.

This work aims to apply this new technique with the primary objective of reducing the progression-free survival for multiple myeloma of patients treated for solitary plasmacytoma, as well as quantify overall survival, local control, toxicities and quality of life in a phase I trial / II.

DETAILED DESCRIPTION:
Solitary plasmacytoma is a rare disease whose treatment has not evolved much in the last decades. The role of radiotherapy in the curative treatment of this entity was defined in a major publication in the 1980s and has since been proven to be the best practice in several other comparative trials, mostly retrospective. The radiotherapy dose of curative intent has also been described over the same period and remains unchanged to this day. Thus, local control, disease cure rate, and rate and progression time for multiple myeloma have been unaffected for almost 30 years.

Radiobiology of plasmacytoma cells is also not widely studied. The alpha / beta ratio, which defines the pattern of response of this disease to radiotherapy fractions and its response time, is also not well described. However, it is believed to be smaller in comparison to other hematological malignancies due to reports of cases of intrinsic radioresistance and late recurrence and reports of success with hypofractionated dose in isolated cases where stereotactic techniques were used such as base of skull and spine.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven plasmacytic for the index lesion;
* Age between 18 and 85 years;
* ECOG scale performance of 0 to 2

Exclusion Criteria:

* Refuse to sign or inability to understand the term of free and informed commitment (TCLE);
* Technical limitations for treatment with SBRT among which is cited, but not limited to, weight greater than 115 Kg, inability to abduct limb to be treated in appendicular bone plasmocytomas, intolerable pain to remain in treatment position;
* Criteria for multiple myeloma at diagnosis: more than 10% of plasma cells in bone marrow biopsy, hypercalcemia greater than 11.5 mg/dL, serum creatinine greater than 2mg/dL, creatinine clearance less than 40mL/min , Hemoglobin less than 10g/dL.
* Previous cancer diagnosis and treatments;
* Previous bone events such as fractures and osteomyelitis in the bone in which the index lesion is found;
* Prior autoimmune diseases, even if controlled;
* Extra-medullary plasmacytoma requiring elective treatment of lymph node drainage;
* Current pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Progression-free survival for multiple myeloma | 5 years
  Progression-free survival for multiple myeloma at 5 years evaluation in patients undergoing SBRT for solitary plasmacytoma compared to a retrospective cohort of patients

SECONDARY OUTCOMES:
Local control rate | 5 years
  Local progression-free survival
Overall survival | 5 years
  Overall survival
Survival free of bone events | 5 Years
  Those are described as fractures, osteomyelitis, necessity of surgery, deformation of bone or ironic bone pain
Toxicities | 5 Years
  Toxicities in the scale of common criteria of toxicity by the National Cancer Institute CTCAE v4
Quality of Life | 5 years
  Quality of life of patients in the prospective cohort using the EORTC QLQ-30 questionnaire
Quality of Life | 5 years
  Quality of life of patients in the prospective cohort using the Short Form Health Survey 36 v.2 (SF-36) questionnaire

OTHER OUTCOMES:
Dosimetric prognostic factors | 5 years
  Describe and explore dosimetric factors for local control and toxicities

CONTACTS AND LOCATIONS:
Locations (1):
- Sao Paulo Cancer Institute, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mill WB, Griffith R. The role of radiation therapy in the management of plasma cell tumors. Cancer. 1980 Feb 15;45(4):647-52. doi: 10.1002/1097-0142(19800215)45:43.0.co;2-e. PMID 6153562
- [Result] Li QW, Niu SQ, Wang HY, Wen G, Li YY, Xia YF, Zhang YJ. Radiotherapy Alone is Associated with Improved Outcomes Over Surgery in the Management of Solitary Plasmacytoma. Asian Pac J Cancer Prev. 2015;16(9):3741-5. doi: 10.7314/apjcp.2015.16.9.3741. PMID 25987031
- [Result] Mendenhall CM, Thar TL, Million RR. Solitary plasmacytoma of bone and soft tissue. Int J Radiat Oncol Biol Phys. 1980 Nov;6(11):1497-501. doi: 10.1016/0360-3016(80)90006-1. No abstract available. PMID 6780494
- [Result] Ozsahin M, Tsang RW, Poortmans P, Belkacemi Y, Bolla M, Dincbas FO, Landmann C, Castelain B, Buijsen J, Curschmann J, Kadish SP, Kowalczyk A, Anacak Y, Hammer J, Nguyen TD, Studer G, Cooper R, Sengoz M, Scandolaro L, Zouhair A. Outcomes and patterns of failure in solitary plasmacytoma: a multicenter Rare Cancer Network study of 258 patients. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):210-7. doi: 10.1016/j.ijrobp.2005.06.039. Epub 2005 Oct 17. PMID 16229966
- [Result] Wong ET, Lu XQ, Devulapalli J, Mahadevan A. Cyberknife radiosurgery for basal skull plasmacytoma. J Neuroimaging. 2006 Oct;16(4):361-3. doi: 10.1111/j.1552-6569.2006.00062.x. PMID 17032388
- [Result] Chang UK, Lee DH, Kim MS. Stereotactic radiosurgery for primary malignant spinal tumors. Neurol Res. 2014 Jun;36(6):597-606. doi: 10.1179/1743132814Y.0000000381. Epub 2014 Apr 28. PMID 24773479
- [Result] Timmerman RD. An overview of hypofractionation and introduction to this issue of seminars in radiation oncology. Semin Radiat Oncol. 2008 Oct;18(4):215-22. doi: 10.1016/j.semradonc.2008.04.001. No abstract available. PMID 18725106